CLINICAL TRIAL: NCT05734027
Title: COMPARISON OF SECTIONAL MATRIX VERSUES CIRCUMFERENTIAL MATRIX FOR RECONSTRUCTION OF PROXIMAL CONTACT IN CLASS 2 RESTORATIONS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Pakistan Institute of Medical Sciences (Other Government)
Responsible Party: Principal Investigator, sheejia asif, Principal investigator, Pakistan Institute of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SOD/ERB/2023/18
Record Dates: First submitted 2023-02-09; First posted 2023-02-17 (Actual); Last update posted 2023-02-17 (Actual); Status verified 2023-02

CONDITIONS: Tooth Decay
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sectional matrix band (Experimental): precontoured sectional matrix band
  Interventions: Device: Sectional matrix; Device: Circumferential matrix
- Circumferential matrix band (Active Comparator): Circumferential matrix band applied by tofflemire retainer
  Interventions: Device: Sectional matrix; Device: Circumferential matrix

INTERVENTIONS:
Device: Sectional matrix — The sectional matrix is the best way to achieve a strong contact point in Class II restorations with composite resin in the posterior dental sector. The pre-wedging is essential to get a separation between teeth which avoid the matrix deformation during its insertion
Device: Circumferential matrix — Circumferential matrix (thickness 0.038mm) ,the band encircle the tooth and secured by retainer on the buccal and lingual aspect

SUMMARY:
Class II caries affects proximal surfaces of premolars and maintain their anatomical proximal contact of tooth, is important to avoid food impaction in the interdental area for protection of periodontium and occurrence of secondary carious lesion.Different types of Matrix band system are used to restore tooth cavities with missing proximal walls, including flat or pre-contoured bands, retainer-fixed circumferential systems, and sectional matrices, and either metal or plastic matrices which produces good contours and contacts for use with amalgam and can also be employed for insertion of composite resin.This study aimed at assessing the influence of different matricing techniques :either sectional matrix or circumferential matrix and the influence of operator experience on reproduction of optimum proximal contacts for posterior proximal resin composite restorations.

DETAILED DESCRIPTION:
Local anesthesia will be administrated, and the whole quadrant containing the offending tooth will be isolated by using a rubber dam.After caries removal and cavity preparation, matrix systems will be applied by dentist ; using either a sectional matrix system and circumferential matrix system.A properly sized wedge will be used with both systems to secure both matrices in place cervically and to prevent gingival overhangs , Resin composite restorations will be completed according to the manufacturer's instructions. Selective enamel etching will be performed by using etchant followed by applying Single Bond Universal adhesive to the entire surface of the enamel and dentin. Then, a thin layer of flowable composite will be applied to ensure adaptation at the gingival margin. Finally, prepared cavities will be restored by using resin composite. using the centripetal technique to build a proximal wall initially followed by successive cusp building. Restorations will be finished by using a flame-shaped finishing stone and polished, and the occlusal contact points will be checked by using a articulating paper. Tightness of proximal contacts will be evaluated using dental floss . For assessment of the restoration, the patients will be sitting in a dental unit with a standardized seating position, which will be reproduced by the unit's preset positioning system, and assessors evaluated the proximal contact by using unwaxed dental floss following theFDI recommendations accordingly to be either optimum, tight, or open contact.Proximal contacts will be categorized as optimum, open, and tight; if the dental floss passed through the contact area as natural dentition on the other side, it will be considered as an optimum contact point. Open contact points will be considered when the dental floss passed through the contact area without resistance; however, when the dental floss could not be passed at all or tore, proximal contact will be considered as tight.

ELIGIBILITY:
Inclusion Criteria:

Tooth with compound class 2 cavities Patient with good general health. Patient with minimum age of 18 years. Fully erupted occluding premolar and molar teeth.

Exclusion Criteria:

Tooth complex class 2 cavities. Tooth with severe periodontal disease. Diastema between posterior teeth. Third molars are excluded.

. Tooth mobility greater than 1 mm.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-08-27 (Actual); Primary Completion 2023-03-02 (Estimated); Study Completion 2023-03-10 (Estimated)

PRIMARY OUTCOMES:
Tightness of proximal contact | immediately after the procedure
  Proximal contact either optimum, tight, or open contact by using dental floss

CONTACTS AND LOCATIONS:
Locations (1):
- Pims ,school of dentistry, Islamabad, Pakistan

IPD SHARING:
Plan to Share IPD: No